CLINICAL TRIAL: NCT06190431
Title: Does the Coaching Function Improve the Learning of Mechanical In-exsufflation (MI-E) in Paediatric Subjects?
Acronym: MI-Ecoaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI-E coaching project
Record Dates: First submitted 2023-12-08; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Cough; Airway Clearance Impairment; Neuromuscular Diseases
Keywords: Mechanical In-Exsufflation; Coaching; Cough Assistance; Pediatric
MeSH Terms: conditions — Cough; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Only physiotherapist guidance (Active Comparator): The aim of this study is to test whether the use of a coaching module (playful visual stimulation) in addition to guidance by a physiotherapist improves the learning and effectiveness of the technique compared to guidance alone.
  Interventions: Other: Learning the use of an in-exsufflation device with the guidance of a physiotherapist
- Physiotherapist guidance + coaching module (Active Comparator): The aim of this study is to test whether the use of a coaching module (playful visual stimulation) in addition to guidance by a physiotherapist improves the learning and effectiveness of the technique compared to guidance alone.
  Interventions: Other: Learning the use of an in-exsufflation device with the guidance of a physiotherapist; Other: Using the coaching mode

INTERVENTIONS:
Other: Learning the use of an in-exsufflation device with the guidance of a physiotherapist — Learning to use an in-exsufflation device with the guidance of a physiotherapist
Other: Using the coaching mode — Learning the use of an in-exsufflation device using a coaching mode (playful visual stimulation) in addition to guidance of a physiotherapist
  Arms: Physiotherapist guidance + coaching module

SUMMARY:
The use of mechanical insufflation-exsufflation (MI-E) in children with neuromuscular diseases (NMD) is recommended by international guidelines and societies and well documented. Many authors have shown that MI-E is safe and effective for airway clearance and has a significant benefit in reducing the duration of the airway clearance session in children with respiratory infections and atelectasis or in the postoperative period. However, its use in paediatrics is still poorly supervised and learning the technique is too often therapist- and/or patient-dependent. The use of a protocol or means of help to guide the initiation and learning of MI-E would allow better use, better adaptation of the settings and potentially better compliance with the treatment. The aim of this study is to test whether the use of a coaching module (playful visual stimulation) in addition to guidance by a physiotherapist improves the learning and effectiveness of the technique compared to guidance alone.This randomized controlled study will first include healthy children, aged 6 to 12 years, with no history or recent respiratory infection affecting lung function or other chronic diseases. In a second phase, the investigators will test the use of the learning process in children with neuromuscular diseases. The investigators hope that the results of this study will provide a better framework for the learning and effectiveness of MI-E. Furthermore, if the results are positive, this will allow better support for the use of MI-E in chronic treatments and help to ensure that this costly treatment for hospitals and public health is used efficiently.

DETAILED DESCRIPTION:
RATIONALE In the first part, the population will be composed of healthy children, in the second part, the investigators will include children with neuromuscular diseases. The two parts will follow the same process. The hypothesis is that the use of a coaching module (playful visual stimulation) in addition to guidance by a physiotherapist improves the learning and effectiveness of the MI-E compared to guidance alone. The MI-E technique does not represent any documented risk in its use nor in its indication if the contraindications are respected (non-drained pneumothorax, hemoptysis and hemodynamic instability). Coaching modules (playful visual stimulation) have recently become available on MI-E devices. This experiment will allow us to judge their usefulness in teaching the use of MI-E in paediatric patients.

OBJECTIVES The aim of this study is to test whether the use of a coaching module (playful visual stimulation) in addition to guidance by a physiotherapist improves the learning and effectiveness of the technique compared to guidance alone. This randomized controlled study will first include healthy children, aged 6 to 12 years. In a second phase, the investigators will test the use in children with neuromuscular diseases. For the process (common for the two parts), eligible subjects will be invited to perform, depending on randomization at the intervention 1 (physiotherapist guidance + coaching module) or the intervention 2 (physiotherapist guidance). The learning times, the coughing expiratory flow rate achieved and the synchronization between the subject and the machine will be compared between the two processes.

ELIGIBILITY:
Part 1:

* Inclusion criteria

  * Age 6-12 (F/M)
  * Acceptance of consent (child + 2 parents)
  * Non-smoker
  * Speak and understand French
  * Schooling in mainstream education
* Exclusion criteria

  * Comorbidities: congenital heart disease, chronic lung disease, immune deficiency, neuromuscular disease, neurological disease or multiple disabilities
  * History or clinical signs of disease affecting lung function, recent lung infection, spinal or thoracic deformity.

Part 2:

* Inclusion criteria

  * Age 6-12 (F/M)
  * Acceptance of consent (child + 2 parents)
  * Non-smoker
  * Speak and understand French
  * Patient with a neuromuscular disease
  * Able to perform the MI-E maneuver
* Exclusion criteria

  * Hemodynamic instability
  * Current or recent pneumothorax
  * Hemoptysis

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | A the end of the learning session (after maximum 15 minutes)
  The investigators will measure the number of sets (n) needed by the subjects to achieve five quality voluntary coughs during the learning session.
Effectiveness | A the end of the learning (after maximum 15 minutes).
  The investigators will measure the time needed (sec) by the subjects to achieve five quality voluntary coughs during the learning session.

SECONDARY OUTCOMES:
Peak cough flow measured with the device (L/min) | During the learning session (max 15 minutes)
  The peak cough flow reached with the In-exsufflation device will be reported
Peak cough flow measured with the device (L/min) | During the session on the second day (24 hours after the learning session)
  The peak cough flow reached with the In-exsufflation device will be reported
Visual analog scales (VAS) "ease of use" (0-10) | At the end of the learning session (max 15 minutes)
  Children will be assessed about the ease of the learning
Visual analog scales (VAS) "ease of use" (0-10) | At the end of the session on the second day (24 hours after the learning session)
  Children will be assessed about the ease of the learning
Visual analog scales (VAS) "comfort" (0-10) | At the end of the learning session (max 15 minutes)
  Children will be assessed about the comfort of the procedure
Visual analog scales (VAS) "comfort" (0-10) | At the end of the session on the second day (24 hours after the learning session)
  Children will be assessed about the comfort of the procedure
the number of sets (n) | At the end of the session on the second day (24 hours after the learning session)
  The investigators will measure the number of sets (n) needed by the subjects to achieve five Quality voluntary coughs one day after the first session.
the time (sec) needed by the subjects to achieve five Quality voluntary coughs | At the end of the session on the second day (24 hours after the learning session)
  The investigators will measure the time (sec) needed by the subjects to achieve five Quality voluntary coughs one day after the learning session.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Audag, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panitch HB. Respiratory Implications of Pediatric Neuromuscular Disease. Respir Care. 2017 Jun;62(6):826-848. doi: 10.4187/respcare.05250. PMID 28546380
- [Background] Miske LJ, McDonough JM, Weiner DJ, Panitch HB. Changes in gastric pressure and volume during mechanical in-exsufflation. Pediatr Pulmonol. 2013 Aug;48(8):824-9. doi: 10.1002/ppul.22671. Epub 2012 Sep 4. PMID 22949331
- [Background] Hov B, Andersen T, Toussaint M, Mikalsen IB, Vollsaeter M, Markussen H, Indrekvam S, Hovland V. User-perceived impact of long-term mechanical assisted cough in paediatric neurodisability. Dev Med Child Neurol. 2023 May;65(5):655-663. doi: 10.1111/dmcn.15543. Epub 2023 Feb 14. PMID 36787316
- [Background] Hull J, Aniapravan R, Chan E, Chatwin M, Forton J, Gallagher J, Gibson N, Gordon J, Hughes I, McCulloch R, Russell RR, Simonds A. British Thoracic Society guideline for respiratory management of children with neuromuscular weakness. Thorax. 2012 Jul;67 Suppl 1:i1-40. doi: 10.1136/thoraxjnl-2012-201964. No abstract available. PMID 22730428
- [Background] Hov B, Andersen T, Toussaint M, Vollsaeter M, Mikalsen IB, Indrekvam S, Hovland V. Prevalence of long-term mechanical insufflation-exsufflation in children with neurological conditions: a population-based study. Dev Med Child Neurol. 2021 May;63(5):537-544. doi: 10.1111/dmcn.14797. Epub 2021 Jan 3. PMID 33393110